CLINICAL TRIAL: NCT02141074
Title: An Open-label Single-arm Multicentre Non-controlled Phase 3 a Trial Investigating Safety and Efficacy of Nonacog Beta Pegol (N9-GP) in Prophylaxis and Treatment of Bleeding Episodes in Previously Untreated Patients With Haemophilia B (FIX Activity Below or Equal to 2 Percent)
Brief Title: Safety and Efficacy of Nonacog Beta Pegol (N9-GP) in Previously Untreated Patients With Haemophilia B
Acronym: paradigm™6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7999-3895; 2012-004867-38 (EudraCT Number); U1111-1135-9557 (Other: WHO); JapicCTI-142611 (Registry Identifier: JAPIC); NL53683.091.15 (Other: CCMO)
Record Dates: First submitted 2014-03-28; First posted 2014-05-19 (Estimated); Results first posted 2023-12-29 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Congenital Bleeding Disorder; Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 50 EDs (exposure days) (Experimental)
  Interventions: Drug: nonacog beta pegol

INTERVENTIONS:
Drug: nonacog beta pegol — For intravenous (i.v.) injection. A single dose of 40 U/kg, unless the bleeding episode is severe in which case it should be treated with 80 U/kg.

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate the safety and efficacy of nonacog beta pegol (N9-GP) in previously untreated patients with Haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male, age below 6 years at the time of signing informed consent
* Patients with the diagnosis of haemophilia B (FIX (coagulation factor IX) activity level below or equal to 2%) based on medical records or central laboratory results
* Previously untreated or exposed to FIX containing products less than or equal to 3 exposure days (5 previous exposures to blood components is acceptable)

Exclusion Criteria:

* Any history of FIX inhibitors (defined by medical records)
* Known or suspected hypersensitivity to trial product or related products
* Previous participation in this trial. Participation is defined as first dose administered of trial product
* Receipt of any investigational medicinal product within 30 days before screening
* Congenital or acquired coagulation disorder other than haemophilia B
* Any chronic disorder or severe disease which, in the opinion of the Investigator, might jeopardise the patient's safety or compliance with the protocol
* Patient's parent(s)/LAR(s) (legally acceptable representative) mental incapacity, unwillingness to cooperate, or a language barrier precluding adequate understanding and cooperation

Ages: 0 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (93):
- United States (23):
  - Miller Children's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Nemours Chld Clnc Jacksonville, Jacksonville, Florida
  - Augusta University, Augusta, Georgia
  - Hope for Kids, Macon, Georgia
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - University Of Iowa, Iowa City, Iowa
  - Children's Hosp-New Orleans, New Orleans, Louisiana
  - Johns Hopkins University_Baltimore_3, Baltimore, Maryland
  - Univ of NE Med Center_Omaha, Omaha, Nebraska
  - North Shore Long Island Jewish Medical Center, New Hyde Park, New York
  - University of North Carlolina-Chapel Hill, Chapel Hill, North Carolina
  - Novant Hlth Vasc Ins Charlotte, Charlotte, North Carolina
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Dayton Children Hemostati Ctr, Dayton, Ohio
  - Penn State MS Hershey Med Ctr, Hershey, Pennsylvania
  - St Christopher Hosp for Child, Philadelphia, Pennsylvania
  - Medical University Of SC, Charleston, South Carolina
  - Vanderbilt Hemostasis Thrombosis Clinic, Nashville, Tennessee
  - Univ of Utah Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - Children's Hsptl Of The Kings, Norfolk, Virginia
- Algeria (2):
  - Beni Messous Hospital Issaad Hassani, Algiers
  - University Hospital Saadna Abdenour of Setif, Sétif
- Argentina (2):
  - Hospital de Pediatría S.A.M.I.C. "Prof. Dr. Juan P. Garrahan, CABA
  - Sanatorio Mayo Privado S.A, Córdoba
- Australia (2):
  - Lady Cilento Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Austria (7):
  - Med. Univ. Graz -Klinische Abteilung f. Allgemeine Pädiatrie, Graz
  - Universitätsklinik Kinder-Jugendheilkunde Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee (LKH Klagenfurt), Klagenfurt
  - Landes-Frauen und Kinderklinik Linz, Linz
  - LKH Salzburg- Univ. Klinik f. Kinder- und Jugendheilkunde, Salzburg
  - Ordination Prof. Zwiauer, Sankt Pölten
  - Universitätsklinik für Kinder- und Jugendheilkunde, Vienna
- UMHAT Sveti Georgi EAD, Plovdiv, Clinic of Pediatrics, Plovdiv, Bulgaria
- Canada (2):
  - Hamltn Hth Sci/McMstr Child Hosp, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- France (5):
  - CHU Estaing, Clermont-Ferrand
  - Ap-Hp-Hopital de Bicetre-1, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Nantes-Hopital Hotel-Dieu, Nantes
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - CHU Haute Pierre, Strasbourg
- Germany (4):
  - Universitätsklinikum Bonn - Institut für Experimentelle Hämatologie, Bonn
  - Coagulation Research Center, Duisburg
  - HZRM Haemophilie-Zentrum Rhein Main GmbH, Frankfurt am Main
  - Werlhof-Institut, Hanover
- Greece (2):
  - Aghia Sophia Childrens' Hospital, Athens
  - 'Ippokrateio' General Hospital of Thessaloniki, Thessaloniki
- Sheba MC - The Israeli National Hemophilia Center, Tel Litwinsky, Israel
- Italy (2):
  - Dipartimento di Ematologia Univ. Firenze, Florence
  - IRCCS Meyer Firenze, Florence
- Japan (6):
  - Nagoya University Hospital_Blood Transfusion, Aichi
  - Kanagawa Children's Medical Center _ Hematology / Oncology, Kanagawa
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
  - Shizuoka Children's Hospital, Hematology-Oncology, Shizuoka
  - National Center for Child Health and Development_Hematology, Tokyo
  - Ogikubo Hospital_Pediatries & Blood, Tokyo
- Malaysia (4):
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - Hospital Pulau Pinang_Georgetown, Penang, George Town, Pulau Pinang
  - Hospital Tengku Ampuan Rahimah, Klang, Selangor
  - National Blood Centre, Kuala Lumpur
- Mexico (2):
  - Centro Medico Nacional SXXI-Hospital de Pediatria, IMSS, Mexico City, México, D.F.
  - Hospital Universitario Dr. José Eleuterio González_Monterrey, Monterrey, Nuevo León
- Radboudumc, Nijmegen, Netherlands
- Portugal (2):
  - Centro Hospitalar Lisboa Norte-HSM, Lisbon
  - ULS São João, E.P.E., Porto
- Romania (2):
  - ,,Louis Ţurcanu'' Emergency Hospital for Children, Timișoara, Timiș County
  - 1st Paediatric Department, Fundeni Clinical Institute, Bucharest
- Serbia (2):
  - University Children's Hospital Tirsova, Belgrade
  - Institute for Mother and Child Health Care of Serbia, Belgrade
- Spain (3):
  - Hospital Sant Joan de Déu, Esplugues Llobregat
  - Hospital Universitario La Paz, Madrid
  - Hospital La Fe - Endocrinología y Nutrición, Valencia
- Taiwan (6):
  - Changhua Christian Hospital_Hematology Dept., Changhua
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital_Dept of Pediatrics, Kaohsiung City
  - China Medical University Children's Hospital, Taichung
  - China Medical University Hospital - Children Building, Taichung
  - National Taiwan University Children's Hospital, Taipei
- Thailand (3):
  - King Chulalongkorn Memorial Hospital_Pediatric Hematology-Oncology, Bangkok
  - Ramathibodi Hospital_Paediatrics, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital _Pediatric Hematology and Oncology, Chiang Mai
- Ukraine (2):
  - SI Institute of Urgent and Recovery Surgery - Haematology, Donetsk
  - Institute of blood pathology and transfusion medicine of NAMSU - General and haematol. surgery, Lviv
- United Kingdom (7):
  - Birmingham Children's Hospital, Birmingham
  - Kent and Canterbury Hospital - Kent Haemophilia and Thrombosis Centre, Canterbury
  - Royal Hospital for Children, Glasgow
  - Leicester Royal Infirmary - Haemostasis & Thrombosis Unit, Leicester
  - St Thomas' Hospital - Haemostasis and Thrombosis Centre, London
  - Royal Manchester Children's Hospital, Manchester
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Background] Chan AK, Alamelu J, Barnes C, Chuansumrit A, Garly ML, Meldgaard RM, Young G. Nonacog beta pegol (N9-GP) in hemophilia B: First report on safety and efficacy in previously untreated and minimally treated patients. Res Pract Thromb Haemost. 2020 Jul 29;4(7):1101-1113. doi: 10.1002/rth2.12412. eCollection 2020 Oct. PMID 33134776
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 29 sites in 11 countries as follows (number of sites that screened participants/ number of sites that randomised participants): Australia (1/1); Austria (2/2); Canada (1/1); Israel (1/1); Japan (1/1); Malaysia (4/4); Spain (3/3); Taiwan (2/2); Thailand (2/2); United Kingdom (3/3); United States (9/9).
Pre-assignment Details: Trial consists of main phase including pre-prophylaxis & prophylaxis, extension phase & prophylaxis period until end of treatment. Pre-prophylaxis was optional and allowed participants to receive treatment until 24 months of age/upon reaching 20EDs, whichever came first. Other participants directly started on prophylaxis treatment at visit 1.
Groups:
- Pre-prophylaxis: Participants received nonacog beta pegol 40 international units/kilogram (IU/kg) intravenous injection at intervals longer than a week on-demand for bleeding episodes until they were 24 months of age or until 20 exposure days (ED), whichever came first, in the main phase. Participants switched from pre-prophylaxis treatment to prophylaxis treatment no later than 24 months of age/20 ED, whichever came first.
- Prophylaxis: Participants who started with pre-prophylaxis were switched to prophylaxis no later than 24 months of age or upon reaching 20EDs, whichever came first. These participants that switched from pre-prophylaxis and other participants who started directly on prophylaxis since visit 1 received once weekly dosing of nonacog beta pegol 40 IU/kg intravenous injection in the main phase, extension phase, and until the end of treatment.
Period: Pre-prophylaxis
Arm/Group | Pre-prophylaxis | Prophylaxis
Started | 34 | 0
Completed | 31 | 0
Not Completed | 3 | 0
Not completed — Adverse Event | 3 | 0
Period: Prophylaxis
Arm/Group | Pre-prophylaxis | Prophylaxis
Started | 0 | 51 (31 participants from Pre-prophylaxis period continued to the Prophylaxis period and additional 20 participants directly started the Prophylaxis period.)
Completed | 0 | 41
Not Completed | 0 | 10
Not completed — Withdrawal by parent/guardian | 0 | 2
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawn due to closure of trial | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set: all participants exposed to study drug. Participants switched from pre-prophylaxis treatment to prophylaxis treatment. Other participants directly started on prophylaxis treatment at visit 1. Pre-prophylaxis and Prophylaxis arms are not mutually exclusive so the data in this section is provided for all participants that started the study.
Groups:
- Nonacog Beta Pegol: Participants received pre-prophylaxis treatment of nonacog beta pegol 40 IU/kg intravenous injection at intervals longer than a week on-demand for bleeding episodes until they were 24 months of age or until 20 exposure days (ED) whichever came first in the main phase. After which they switched to prophylaxis treatment. In prophylaxis, participants received nonacog beta pegol 40 IU/kg intravenous injection once weekly in the main phase, extension phase and until end of treatment.
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.8 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 19
  Black or African American | 7
  White | 25
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Inhibitory Antibodies Against Coagulation Factor IX (FIX) (50 Exposure Days)
Description: Number of participants with incidence of inihibitory antibodies against FIX after 50 ED is presented and defined as an inhibitory antibody titre greater than equal to 0.6 Bethesda unit (BU) at two consecutive tests performed at the central laboratory and also tested positive for nonacog beta pegol binding antibodies.
Time Frame: When minimum 20 previously untreated patients (PUPs) have reached at least 50 exposure days (ED) (up to 156 weeks)
Population: Safety analysis set included all participants exposed to nonacog beta pegol. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 28
Participants | 2 | 0

2. Primary Outcome: Number of Participants With Incidence of Inhibitory Antibodies Against FIX (100 ED)
Description: Number of participants with incidence of inihibitory antibodies against FIX after 100 ED is presented and defined as an inhibitory antibody titre greater than equal to 0.6 Bethesda unit (BU) at two consecutive tests performed at the central laboratory and also tested positive for nonacog beta pegol binding antibodies.
Time Frame: When minimum 40 PUPs have reached at least 100 ED (up to 208 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 19 | 47
Participants | 2 | 2

3. Primary Outcome: Number of Participants With Incidence of Inhibitory Antibodies Against FIX (At End of Trial)
Description: Number of participants with incidence of inihibitory antibodies against FIX at end of trial is presented and defined as an inhibitory antibody titre greater than equal to 0.6 Bethesda unit (BU) at two consecutive tests performed at the central laboratory and also tested positive for nonacog beta pegol binding antibodies.
Time Frame: At end of trial (up to 434 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 20 | 51
Participants | 2 | 2

4. Secondary Outcome: Number of Adverse Events
Description: Number of adverse events after 50 ED, after 100 ED, and at end of trial is presented. An adverse event was defined as any untoward medical occurrence in a participant who was administered a product, and which does not necessarily have a causal relationship with this treatment. All presented adverse events are treatment emergent adverse events, defined as an event that occured while the participant was on treatment in the period from first dosing with nonacog beta pegol to the end of trial/discontinuation of treatment.
Time Frame: When minimum 20 PUPs have reached at least 50 ED (up to 156 weeks); when minimum 40 PUPs have reached at least 100 ED (up to 208 weeks); at end of trial (up to 434 weeks)
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Events
  50 ED: number analyzed (Participants) | 24 | 28
  50 ED | 86 | 291
  100 ED: number analyzed (Participants) | 32 | 47
  100 ED | 131 | 610
  End of trial (Week 434) | 134 | 794

5. Secondary Outcome: Frequency of Adverse Events
Description: Frequency of adverse events after 50 ED, after 100 ED, and at end of trial is presented. Frequency of adverse events was expressed as number of adverse events per participant years of exposure (total number of events /total time in trial). An adverse event was defined as any untoward medical occurrence in a participant who was administered a product, and which does not necessarily have a causal relationship with this treatment. All presented adverse events are treatment emergent adverse events, defined as an event that occured while the participant was on treatment in the period from first dosing with nonacog beta pegol to the end of trial/discontinuation of treatment.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Events per participant years of exposure
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Events per participant years of exposure
  50 ED: number analyzed (Participants) | 24 | 28
  50 ED | 5.59 | 5.87
  100 ED: number analyzed (Participants) | 32 | 47
  100 ED | 5.92 | 5.08
  End of trial (Week 434) | 5.52 | 4.10

6. Secondary Outcome: Number of Serious Adverse Events
Description: Number of serious adverse events after 50 ED, after 100 ED, and at end of trial is presented. A serious adverse event was an experience that at any dose resulted in: death; life-threatening experience; in-patient hospitalisation or prolongation of existing hospitalisation; a persistent or significant disability/incapacity; congenital anomaly/birth defect; important medical events that may not result in death, be life-threatening/require hospitalisation could be considered a serious adverse event based upon appropriate medical judgement.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Events
  50 ED: number analyzed (Participants) | 24 | 28
  50 ED | 9 | 14
  100 ED: number analyzed (Participants) | 32 | 47
  100 ED | 13 | 27
  End of trial (Week 434) | 14 | 30

7. Secondary Outcome: Frequency of Serious Adverse Events
Description: Frequency of serious adverse events after 50 ED, after 100 ED, and at end of trial is presented. Frequency of serious adverse events was expressed as number of serious adverse events per participant years of exposure (total number of events /total time in trial). A serious adverse event was an experience that at any dose resulted in: death; life-threatening experience; in-patient hospitalisation or prolongation of existing hospitalisation; a persistent or significant disability/incapacity; congenital anomaly/birth defect; important medical events that may not result in death, be life-threatening/require hospitalisation could be considered a serious adverse event based upon appropriate medical judgement.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Events per participant years of exposure
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Events per participant years of exposure
  50 ED: number analyzed (Participants) | 24 | 28
  50 ED | 0.59 | 0.28
  100 ED: number analyzed (Participants) | 32 | 47
  100 ED | 0.59 | 0.22
  End of trial (Week 434) | 0.58 | 0.15

8. Secondary Outcome: Number of Medical Events of Special Interest
Description: Number of medical events of special interest after 50 ED, after 100 ED, and at end of trial is presented. A medical event of special interest (MESI) was an event that, in the evaluation of safety, has a special focus. A MESI was an adverse event (serious or non-serious adverse event) that fulfils one or more of the following MESI criteria: 1. Medication errors concerning the trial product; 2. Inhibitor formation against FIX; 3. Thromboembolic events; 4. Anaphylactic reaction; 5. Allergic reaction including, but not limited to, any acute immunoglobulin E mediated reaction of delayed-type hypersensitivity (clinical signs may include various types of skin rashes) that does not meet the definition of anaphylaxis; 6. CNS-related adverse events including, but not limited to, any learning and behavioral deficits; 7. Renal adverse events including new onset of renal disorder or renal impairment or acute and chronic renal failure.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Events
  50 ED: number analyzed (Participants) | 24 | 28
  50 ED | 5 | 9
  100 ED: number analyzed (Participants) | 32 | 47
  100 ED | 6 | 31
  End of trial (Week 434) | 6 | 38

9. Secondary Outcome: Frequency of Medical Events of Special Interest
Description: Frequency of medical events of special interest after 50 ED, after 100 ED, and at end of trial is presented. It was expressed as number of MESI per participant years of exposure (total number of events/total time in trial). A MESI was an event that, in the evaluation of safety, has a special focus. A MESI was an adverse event that fulfils one or more of the MESI criteria: 1. Medication errors concerning the trial product; 2. Inhibitor formation against FIX; 3. Thromboembolic events; 4. Anaphylactic reaction; 5. Allergic reaction including, but not limited to, any acute immunoglobulin E mediated reaction of delayed-type hypersensitivity (clinical signs may include various types of skin rashes) that does not meet the definition of anaphylaxis; 6. CNS-related adverse events including, but not limited to, any learning and behavioral deficits; 7. Renal adverse events including new onset of renal disorder or renal impairment or acute and chronic renal failure.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Events per participant years of exposure
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Events per participant years of exposure
  50 ED: number analyzed (Participants) | 24 | 28
  50 ED | 0.33 | 0.18
  100 ED: number analyzed (Participants) | 32 | 47
  100 ED | 0.27 | 0.26
  End of trial (Week 434) | 0.25 | 0.20

10. Secondary Outcome: Number of Breakthrough Bleeding Episodes During Prophylaxis (Annualised Bleeding Rate)
Description: Number of breakthrough bleeding episodes during prophylaxis (annualised bleeding rate) after 50 ED, after 100 ED, and at end of trial is presented. Annualised bleeding rate is the number of bleeding episodes per year.
Time Frame: as for outcome 4
Population: Full analysis set included all participants exposed to nonacog beta pegol. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Median (Full Range); unit: bleeds/participant/year
Units Other Than Participants: bleeding episodes
Arm/Group | Prophylaxis
Number analyzed (Participants) | 51
Number analyzed (bleeding episodes) | 137
bleeds/participant/year
  50 ED: number analyzed (Participants) | 28
  50 ED: number analyzed (bleeding episodes) | 15
  50 ED | 0.00 [0.00 to 2.60]
  100 ED: number analyzed (Participants) | 47
  100 ED: number analyzed (bleeding episodes) | 78
  100 ED | 0.25 [0.00 to 17.39]
  End of trial (Week 434) | 0.33 [0.00 to 17.39]

11. Secondary Outcome: Haemostatic Effect of Nonacog Beta Pegol in Treatment of Bleeding Episodes by 4-point Haemostatic Response Scale ("Excellent", "Good", "Moderate" and "Poor")
Description: Haemostatic effect of nonacog beta pegol in treatment of bleeding episodes by 4-point haemostatic response scale after 50 ED, after 100 ED, and at end of trial is presented. The haemostatic response after treatment of a bleed with nonacog beta pegol was evaluated on a 4-point scale as excellent, good, moderate or poor. Excellent: abrupt pain relief and/or clear improvement in objective signs of bleeding; Good: noticeable pain relief and/or improvement in signs of bleeding; Moderate: probable or slight beneficial effect after the first injection; Poor: no improvement or worsening of symptoms. If the haemostatic response was rated as excellent or good, the treatment of the bleed was considered a success. If the haemostatic response was rated as moderate or poor, the treatment was considered a failure.
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Number; unit: Number of bleeds treated
Units Other Than Participants: Bleeding episodes
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Number analyzed (Bleeding episodes) | 65 | 135
Number of bleeds treated
  50 ED Excellent: number analyzed (Participants) | 24 | 28
  50 ED Excellent: number analyzed (Bleeding episodes) | 33 | 15
  50 ED Excellent | 23 | 9
  50 ED Good: number analyzed (Participants) | 24 | 28
  50 ED Good: number analyzed (Bleeding episodes) | 33 | 15
  50 ED Good | 8 | 5
  50 ED Moderate: number analyzed (Participants) | 24 | 28
  50 ED Moderate: number analyzed (Bleeding episodes) | 33 | 15
  50 ED Moderate | 2 | 1
  50 ED Poor: number analyzed (Participants) | 24 | 28
  50 ED Poor: number analyzed (Bleeding episodes) | 33 | 15
  50 ED Poor | 0 | 0
  100 ED Excellent: number analyzed (Participants) | 32 | 47
  100 ED Excellent: number analyzed (Bleeding episodes) | 63 | 77
  100 ED Excellent | 44 | 44
  100 ED Good: number analyzed (Participants) | 32 | 47
  100 ED Good: number analyzed (Bleeding episodes) | 63 | 77
  100 ED Good | 17 | 30
  100 ED Moderate: number analyzed (Participants) | 32 | 47
  100 ED Moderate: number analyzed (Bleeding episodes) | 63 | 77
  100 ED Moderate | 2 | 3
  100 ED Poor: number analyzed (Participants) | 32 | 47
  100 ED Poor: number analyzed (Bleeding episodes) | 63 | 77
  100 ED Poor | 0 | 0
  End of trial (Week 434) Excellent | 45 | 86
  End of trial (Week 434) Good | 18 | 45
  End of trial (Week 434) Moderate | 2 | 4
  End of trial (Week 434) Poor | 0 | 0

12. Secondary Outcome: Incremental Recovery at 30 Minutes (IR30min)
Description: Incremental recovery 30 minutes post dosing (IR30min) after 50 ED, after 100 ED is presented. IR30min was defined as the rise in FIX activity per international units per kilogram (IU/kg) administered and was recorded 30 minutes after the end of nonacog beta pegol injection. It was calculated as the baseline adjusted FIX activity recorded 30 minutes after ended nonacog beta pegol injection divided by the administered dose (IU/kg body weight). It was recorded as international units per milliliter (IU/mL)/international units per kilogram (IU/kg).
Time Frame: When minimum 20 PUPs have reached at least 50 ED (up to 156 weeks); when minimum 40 PUPs have reached at least 100 ED (up to 208 weeks)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (IU/mL)/(IU/kg)
Arm/Group | Prophylaxis
Number analyzed (Participants) | 25
(IU/mL)/(IU/kg)
  50 ED: number analyzed (Participants) | 14
  50 ED | 0.012 (13.9)
  100 ED | 0.014 (20.1)

13. Secondary Outcome: FIX Activity at 30 Minutes (C30min)
Description: FIX Activity 30 minutes post dosing (C30min) after 50 ED, after 100 ED is presented. The FIX activity was measured by one-stage clotting assay - a modified activated partial thromboplastin time (aPTT) assay.
Time Frame: as for outcome 12
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Prophylaxis
Number analyzed (Participants) | 23
IU/mL
  50 ED: number analyzed (Participants) | 16
  50 ED | 0.652 (39.5)
  100 ED | 0.824 (21.6)

14. Secondary Outcome: FIX Trough Levels
Description: FIX trough levels after 50 ED, after 100 ED, and at end of trial is presented. FIX trough level was defined as the activity recorded immediately before nonacog beta pegol injection was given and was measured by one-stage clotting assay - a modified activated partial thromboplastin time (aPTT) assay. The analysis is based on a mixed model on the log-transformed plasma concentrations with participant as a random effect. The mean trough level is presented back-transformed to the natural scale.
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Prophylaxis
Number analyzed (Participants) | 51
IU/mL
  50 ED: number analyzed (Participants) | 28
  50 ED | 0.150 [0.141 to 0.160]
  100 ED: number analyzed (Participants) | 47
  100 ED | 0.156 [0.144 to 0.170]
  End of trial (Week 434) | 0.167 [0.155 to 0.179]

15. Secondary Outcome: Amount of Drug Administered to Treat a Bleeding Episode
Description: Amount of nonacog beta pegol administered (average dose of nonacog beta pegol) to treat a bleeding episode after 50 ED, after 100 ED, and at end of trial is presented as international units per kilogram per bleed (IU/kg/bleed).
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: IU/kg/bleed
Units Other Than Participants: Bleeding episodes
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Number analyzed (Bleeding episodes) | 65 | 135
IU/kg/bleed
  50 ED: number analyzed (Participants) | 24 | 28
  50 ED: number analyzed (Bleeding episodes) | 33 | 15
  50 ED | 55.0 (28.7) | 48.8 (16.9)
  100 ED: number analyzed (Participants) | 32 | 47
  100 ED: number analyzed (Bleeding episodes) | 63 | 77
  100 ED | 47.7 (17.6) | 58.5 (70.0)
  End of trial (Week 434) | 47.5 (17.4) | 54.0 (53.5)

16. Secondary Outcome: Number of Injections Needed to Treat a Bleeding Episode
Description: The mean number of injections needed to treat a bleeding episode is presented.
Time Frame: as for outcome 4
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Injections per bleed
Units Other Than Participants: Bleeding episodes
Arm/Group | Pre-prophylaxis | Prophylaxis
Number analyzed (Participants) | 34 | 51
Number analyzed (Bleeding episodes) | 65 | 135
Injections per bleed
  50 ED: number analyzed (Participants) | 24 | 28
  50 ED: number analyzed (Bleeding episodes) | 33 | 15
  50 ED | 1.3 (0.7) | 1.0 (0.0)
  100 ED: number analyzed (Participants) | 32 | 47
  100 ED: number analyzed (Bleeding episodes) | 63 | 77
  100 ED | 1.1 (0.4) | 1.3 (1.5)
  End of trial (Week 434) | 1.1 (0.4) | 1.2 (1.2)

ADVERSE EVENTS:
Time Frame: Up to Week 434
Description: All presented adverse events are treatment emergent adverse events, defined as an event that occured while the participant was on treatment in the period from first dosing with nonacog beta pegol to the end of trial/discontinuation of treatment. Safety analysis set included all participants exposed to nonacog beta pegol.
Arm/Group | Pre-prophylaxis | Prophylaxis
All-Cause Mortality (participants affected / at risk) | 1/34 | 1/51
Serious Adverse Events (participants affected / at risk) | 9/34 | 19/51
Other Adverse Events (participants affected / at risk) | 22/34 | 46/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-prophylaxis (N=34) | Prophylaxis (N=51)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Factor IX inhibition (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Language disorder (Nervous system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media viral (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Platelet dysfunction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4)
Poor venous access (Vascular disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-prophylaxis (N=34) | Prophylaxis (N=51)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 6 (7)
Bronchitis (Infections and infestations) | 1 (1) | 6 (8)
COVID-19 (Infections and infestations) | 0 (0) | 6 (7)
Conjunctivitis (Infections and infestations) | 1 (1) | 4 (6)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (8)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 6 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 17 (34)
Dental caries (Gastrointestinal disorders) | 0 (0) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 11 (13)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 4 (5)
Ear infection (Infections and infestations) | 3 (4) | 9 (13)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 8 (14)
Gastroenteritis (Infections and infestations) | 0 (0) | 4 (4)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 4 (4)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 7 (10)
Headache (Nervous system disorders) | 0 (0) | 3 (11)
Influenza (Infections and infestations) | 0 (0) | 5 (6)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (16)
Nasopharyngitis (Infections and infestations) | 5 (12) | 23 (68)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (8)
Otitis media (Infections and infestations) | 2 (2) | 6 (12)
Otitis media acute (Infections and infestations) | 2 (4) | 5 (5)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 11 (23) | 27 (74)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (14)
Rhinitis (Infections and infestations) | 0 (0) | 3 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 9 (21)
Sinusitis (Infections and infestations) | 0 (0) | 3 (5)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 4 (9)
Speech disorder developmental (Nervous system disorders) | 0 (0) | 5 (5)
Teething (Gastrointestinal disorders) | 1 (3) | 4 (7)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tonsillitis (Infections and infestations) | 1 (1) | 5 (8)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 19 (33)
Viral infection (Infections and infestations) | 3 (3) | 5 (10)
Vomiting (Gastrointestinal disorders) | 2 (2) | 11 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT02141074/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02141074/SAP_001.pdf